CLINICAL TRIAL: NCT06387849
Title: Effect of Aromatherapy Using Lavender Essential Oil on Pain and Anxiety After C-section: a Randomized Controlled Trial
Brief Title: Aromatherapy Effect on Pain and Anxiety After C-section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Nesrine Souayeh, Associated Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03/2023
Record Dates: First submitted 2024-04-20; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Post-operative Pain; Post-operative Anxiety
Keywords: Cesarean; Pain; Anxiety; Aromatherapy; Lavender
MeSH Terms: conditions — Pain, Postoperative; Pain; Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy group (Experimental): Two to twelve hours after undergoing C-section, the women enrolled in the experimental arm benefited from aromatherapy with lavender essential oil (EO): The patients were invited to inhale cotton balls, soaked separately with three drops of the EO at a distance of 10 centimeters for 30 minutes.
  Interventions: Other: Aromatherapy
- Placebo (Placebo Comparator): Two to twelve hours after undergoing C-section, the women enrolled in the placebo arm were invited to inhale cotton balls, soaked separately with three drops of the distilled water at a distance of 10 centimeters for 30 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — women enrolled in the experimental group received aromatherapy with lavender essential oil (EO) through dry inhalation (inhalation via a cotton support soaked in a few drops of EO)
  Arms: Aromatherapy group
Other: Placebo — women enrolled in the placebo group received ihaled a cotton support soaked in a few drops of distilled water
  Arms: Placebo

SUMMARY:
A prospective randomized triple blinded study conducted in the obstetrics gynecology department of Ben Arous hospital over a period of four months and 10 days between April 2023 and August 2023.

The aim of this study was to evaluate the effectiveness of lavender aromatherapy on postoperative pain and anxiety after cesarean section under spinal anesthesia in Tunisian women.

ELIGIBILITY:
Inclusion Criteria:

* All women who gave birth by cesarean section under spinal anesthesia in the obstetrics and gynecology department at the Ben Arous regional hospital who met the following criteria were included in this study:

  * Age between 18 and 45 years old
  * Term of pregnancy at the time of delivery ≥ 37 weeks of Gestation.
  * A minimum level of primary education as a prerequisite to answer the questions (in particular the STAI items).
  * Classified ASA 1 or 2 of the American Society of Anesthesiology (ASA) classification.
  * Having no history of cancer or chronic pain.
  * Free from any psychiatric pathology.
  * And having not presented any intra- or post-operative complications.

Exclusion Criteria:

The investigators excluded patients in our study:

* Having given birth to a stillborn or a suffering newborn requiring transfer to neonatal intensive care.
* Having received painkillers in the post-operative period.
* Having olfactory disorders.
* Having a substance abuse problem.
* Having a known allergy to lavender or other aromatic plants.
* who did not agree to participate in the study or who did not continue all stages of the trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pain level | two to twelve hours after surgery
  the investigator evaluated the Post-operative pain level using Visual analogue scale( patient at rest and after ambulation). The score ranges from 0 (no pain at all) to 10 (the worst imaginable pain). the higher the score is, the worst the outcome is.
Post-operative anxiety level | two to twelve hours after surgery
  the investigator evaluated the Post-operative anxiety level using the " State Trait Anxiety Inventory (STAI)forme Y ". The score ranges from 20 to 80. Higher scores are associated with higher levels of anxiety (worse outcome)

SECONDARY OUTCOMES:
Heart Rate (HR) | two to twelve hours after surgery
  Heart Rate in beat per minute (bpm),
Systolic Blood Pressure (SBP) | two to twelve hours after surgery
  Systolic Blood Pressure (SBP) in millimetres of mercury (mmHg)
Diastolic Blood Pressure (DBP) | two to twelve hours after surgery
  Diastolic Blood Pressure (DBP) in millimetres of mercury (mmHg)
Respiratory Rate (RR) | two to twelve hours after surgery
  Respiratory Rate (RR) in cycle per minute (cpm)
Pulsatile Oxygen Saturation | two to twelve hours after surgery
  Pulsatile Oxygen Saturation (SPO2) in percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Hajer Bettaieb, Professor, Study Director — University of Tunis el Manar, Faculty of medicine
Locations (1):
- Ben Arous Regional Hospital, Ben Arous, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nouira M, Souayeh N, Kanzari SA, Rouis H, Lika A, Mbarki C, Rahali FZ, Bettaieb H. Aromatherapy Using Lavender Oil Effectiveness on Pain and Anxiety After C-Section: A Randomized Controlled Trial. J Epidemiol Glob Health. 2024 Dec;14(4):1536-1544. doi: 10.1007/s44197-024-00305-6. Epub 2024 Oct 14. PMID 39400653